CLINICAL TRIAL: NCT07014241
Title: Feasibility Study of Telehealth Family Psychoeducation for Major Depressive Disorder
Brief Title: Assessment of Whether Telehealth Family Psychoeducation for Major Depressive Disorder is Doable
Acronym: SPARKED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Queensland (Other)
Responsible Party: Principal Investigator, Professor Benjamin Tan BNSc MMed PhD RN, Professor of Nursing, University of Southern Queensland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HREC 2025-5059
Record Dates: First submitted 2025-05-26; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Family psychoeducation; Major depressive disorder; Telehealth; Feasibility study
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telehealth family psychoeducation (Experimental): Dyads of individuals with MDD who have been prescribed at least one antidepressant medication and their family members or caregivers
  Interventions: Other: Family psychoeducation

INTERVENTIONS:
Other: Family psychoeducation — The study intervention, tagged SPARKED (Supportive Program for Advancing Recovery, Knowledge, and Empowerment in Depression), is a co-designed family-based psychoeducational intervention for individuals with MDD and their family members or caregivers. The intervention will cover structured modules to enhance participants' understanding of MDD and its treatment, coping strategies, and self-efficacy skills. It will also focus on recognising early signs of relapse and empowering participants to engage actively in treatment decision-making.

SUMMARY:
The goal of this single-arm interventional study is to assess the feasibility and acceptability of co-designed telehealth family psychoeducation (FPE) among individuals with major depressive disorder (MDD) and families. The study will also assess the intervention's preliminary impact on personal recovery, antidepressant medication adherence, depression severity, and medication necessity beliefs and concerns. The main questions it aims to answer are:

* What are patients', families', and mental health professionals' views about telehealth FPE for MDD?
* What are the feasibility and acceptability of telehealth FPE for MDD among individuals with MDD and their families?
* What is the preliminary impact of telehealth FPE for MDD on personal recovery, antidepressant medication adherence, depression severity, and medication necessity beliefs and concerns?

Study participants will include individuals with MDD who have prescriptions for antidepressant medications and their family members. Participants will receive three biweekly FPE sessions and a six-week follow-up session via telehealth using a single-family format. The study intervention, telehealth family psychoeducation for MDD, will cover structured modules to enhance participants' understanding of MDD and its treatment, coping strategies, and self-efficacy skills. It will also focus on recognising early signs of relapse and empowering participants to engage in treatment decision-making actively. Hence, the study intervention is termed the Supportive Program for Advancing Recovery, Knowledge, and Empowerment in Depression (SPARKED).

At baseline, post-intervention, and follow-up, participants with MDD will complete self-reported measures for personal recovery, antidepressant medication adherence, depression severity, and medication necessity beliefs and concerns. In contrast, their family members or caregivers will complete only an outcome measure for medication necessity beliefs and concerns.

ELIGIBILITY:
Inclusion Criteria:

* An individual (aged 18 years or older) with a diagnosis of MDD who has a prescription for at least one antidepressant medication for treating MDD
* The individual has a family member, family caregiver, or significant other (aged 18 years or older) who plays a role in supporting the individual at home
* Both the individual with MDD and their support person have basic English language skills, enabling them to engage in family psychoeducational sessions and respond to self-report outcome measures.
* Both the individual with MDD and their support person voluntarily consent to participate in the study.

Exclusion Criteria:

* An individual (aged 18 years or older) who does not have a prescription for at least one antidepressant medication for treating MDD
* An individual (aged 18 years or older) with MDD whose family member, caregiver, or significant other could not participate in the study
* An individual (aged 18 years or older) with MDD who has high or imminent suicide risk
* An individual with MDD who has other serious mental or physical illnesses, cognitive impairment, or hearing impairment without a hearing aid
* A family member, caregiver, or significant other to an individual with MDD who does not consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Three months beginning on the date the feasibility study flyer is displayed.
  The total number of eligible participant dyads (an individual with MDD and a supportive family member) enrolled on the feasibility study within the recruitment period.
Retention | Across the entire trial period, from enrolment to six-week follow-up.
  The percentage of participants who remain in the study.
Outcome measure return rate | From enrolment to the end of six-week follow-up.
  The percentage of participants who return filled-out self-report measures.
Outcome measure completion rate | From enrolment to the end of the six-week follow-up.
  The percentage of participants who successfully complete a specific outcome measurement.
Prospective acceptability | During the recruitment period, lasting approximately three months.
  Number of eligible participants who consented to study participation
Concurrent acceptability | From the first biweekly session to the end of the six-week follow-up
  Number of family psychoeducational sessions attended and reasons for dropout
Retrospective acceptability. | At six-week follow-up.
  Feedback on telehealth family psychoeducation for MDD, including what worked well, barriers encountered, and suggestions for improvement.

SECONDARY OUTCOMES:
Personal recovery among study participants with MDD | At baseline (T0), immediately post-intervention (T1), and 6-week follow-up (T2)
  This outcome refers to subjective recovery, which will be assessed using the Recovery Assessment Scale-Domains and Stages (RAS-DS), a 38-item self-rated measure of personal recovery.
  The RAS-DS is a 4-point Likert scale that includes four recovery domains: Doing Things I Value, Looking Forward, Mastering My Illness, and Connecting and Belonging. Each item can be rated as "Untrue," "A bit True," "Mostly True," or "Completely True," with corresponding numerical values of 1 to 4. Scores are summed to obtain the total recovery score, with minimum and maximum scores of 38 and 152, respectively. A lower total recovery score suggests a reduced sense of recovery, while a higher score indicates a greater sense of recovery.
  The percentage domain score will be calculated to assess differences across domains at a specific time point and to evaluate changes in the domains over the three measurement time points. Item scores within each domain are summed to obtain the total domain score.
Depressive symptoms among participants with MDD | At baseline (T0), immediately post-intervention (T1), and 6-week follow-up (T2).
  The Patient Health Questionnaire-9 scale, a brief instrument comprising nine items, will be used to evaluate the presence and severity of depressive symptoms. Each item on this scale is rated from 0 to 3, where a score of 0 indicates "Not at all," 1 indicates "Several days," 2 indicates "More than half the days," and 3 indicates "Nearly every day." All scores are summed to get a total score that indicates the severity of depression. The minimum and maximum values are 0 and 27, respectively. A total score of 1-4 indicates minimal depression, 5-9 indicates mild depression, 10-14 indicates moderate depression, 15-19 indicates moderately severe depression, and 20-27 indicates severe depression.
Antidepressant medication adherence among participants with MDD | At baseline (T0), immediately post-intervention (T1), and 6-week follow-up (T2)
  In this study, antidepressant medication adherence refers to how much a person's medication-taking behaviours correspond with a prescriber's recommendations. The medication adherence measurement will involve the Medication Adherence Report Scale-5 (MARS-5), a validated, five-item, self-report measure examining intentional and nonintentional nonadherence behaviours.
  Each item is rated "Always," "Often," "Sometimes," "Rarely," or "Never," which are scored from 1 to 5, respectively. All scores are added up to get a total score. The minimum and maximum values are 5 and 25, respectively. Lower total scores mean lower adherence, while higher total scores indicate higher adherence.
Medication necessity beliefs and concerns among participants with MDD and their family members | At baseline (T0), immediately post-intervention (T1), and 6-week follow-up (T2)
  Necessity beliefs and concerns regarding antidepressant medication will be assessed in all participants using the Beliefs about Medicines Questionnaire-Specific (BMQ-Specific). The BMQ-Specific is an 11-item measure comprising two subscales assessing beliefs about the need for medication prescribed for treatment (Specific-Necessity, five items) and concerns about the medication's potential adverse effects (Specific-Concerns, 6 items).
  Each item is rated as "Strongly Agree," "Agree," "Uncertain," "Disagree," or "Strongly Disagree," and scored from 5 to 1, respectively. Scores on the Specific Necessity scale are summed. Similarly, scores on the Specific Concerns scale are added up. A scale score is determined by dividing the sum of scores on each scale by the respective number of items on the scale. High Specific Necessity scale scores mean strong beliefs about the need for prescribed medication, while high Specific Concerns scale scores mean strong concerns regarding the medications.

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Bakewell Medical Centre, Bakewell, Northern Territory
  - Palmerston Medical Clinic, Palmerston, Northern Territory

IPD SHARING:
Plan to Share IPD: No
The study datasets contain sensitive personal information and are stored securely with restricted access. Access is subject to approval by the relevant ethics committees and data custodians.

REFERENCES:
- [Derived] Obieche O, Tan JB, Sharma S, Bressington D, Wang T. Telehealth Family Psychoeducation for Major Depressive Disorder: A Protocol for Intervention Co-Design and Feasibility Study. Nurs Rep. 2025 Oct 11;15(10):364. doi: 10.3390/nursrep15100364. PMID 41149679